CLINICAL TRIAL: NCT06597591
Title: Acceptability of a VR-based Training for Inhibitory Control in Subjects With Neurocognitive Disorders
Brief Title: Virtual Reality Training for Inhibitory Control in Neurocognitive Disorders
Acronym: VR4IC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-PP-06 VR4IC; Numéro ID RCB: 2024-A01142-45 (Other: ANSM)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Disorder
Keywords: inhibitory control; serious game; virtual reality; cognitive disorder
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: Pseudo-randomisation (controlling for demographic and clinical features, and previous VR experience)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Serious game on VR headset ( immersive VR) (Experimental): After enrolment, patients will have 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game with a VR Headset.
  Interventions: Device: VR headset
- Serious game on tablet ( non Immersive VR) (Experimental): After enrolment, patients will have 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game on a tablet.
  Interventions: Device: Tablet
- Waiting Serious game on VR headset (Waiting immersive VR) (Experimental): 2-month after enrolment, patients will have 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game with a VR Headset.
  Interventions: Device: VR headset
- Waiting Serious game on tablet ( Waiting non Immersive VR) (Experimental): 2-month after enrolment, patients will have 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game with a VR Headset.
  Interventions: Device: Tablet

INTERVENTIONS:
Device: VR headset — 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game with a VR Headset. The serious game is inspired by the GoNoGo task.The players' task is to throw objects in a basket matching the active rule. These objects can be of three different colors (red, yellow, and purple) with the presence or absence of stains on them. The objects' color is hidden until the player interacts with them. Example of rule: the active rule is to throw in the basket only the objects in red without stains, yellow with stains, and purple with stains. To earn points, the player must match the rule presented and throw the objects away if they do not match.
  Arms: Serious game on VR headset ( immersive VR); Waiting Serious game on VR headset (Waiting immersive VR)
Device: Tablet — 8 sessions (2 times per week for 4 weeks) of 20 minutes playing the serious game with a tablet. The serious game is inspired by the GoNoGo task.The players' task is to throw objects in a basket matching the active rule. These objects can be of three different colors (red, yellow, and purple) with the presence or absence of stains on them. The objects' color is hidden until the player interacts with them. Example of rule: the active rule is to throw in the basket only the objects in red without stains, yellow with stains, and purple with stains. To earn points, the player must match the rule presented and throw the objects away if they do not match.
  Arms: Serious game on tablet ( non Immersive VR); Waiting Serious game on tablet ( Waiting non Immersive VR)

SUMMARY:
Executive function disorders, such as inhibitory control (IC) difficulties, are very common in older adults with neurocognitive disorders (NCD). Management of these disorders is possible using traditional tools and tools based on new technologies, such as serious games and virtual reality (VR). However, today, few immersive tools exist that are specifically focused on IC training. The present study aims to evaluate the acceptability of an immersive application focused on IC in 48 patients with neurocognitive disorders. Participants that will test either an immersive (VR-headset) or a non-immersive (tablet) version of the application for 4 weeks, twice a week, and fill-in acceptability related questionnaires before, during and after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. consulting the Nice hospital Memory Center
2. diagnosis of Mild Neurocognitve Disorder or slight major neurocognitive disorder (DSM V)
3. 60 years old or more
4. presence of deficits in inhibitory control as assessed by the Frontal Assessment Battery
5. fluent in French
6. able to understand the informed consent form and voluntarily consents to participate

Exclusion Criteria:

1. presence of significant vision or motor problems which would impact ability to perform the task
2. significant self-reported motion sickness
3. vulnerable persons as defined in articles L1121-5 to 8 of the French Public Health Code

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-05-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Unified Theory of Acceptance and Use of Technology 2 (UTAUT2) Questionnaire | at inclusion
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions..
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.
UTAUT 2 Questionnaire | at 4-week
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions.
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.
UTAUT 2 Questionnaire | at 8-week
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions..
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.
UTAUT 2 Questionnaire | at 16-week
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions..
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.
UTAUT 2 Questionnaire | at 20-week
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions..
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.
UTAUT 2 Questionnaire | at 24-week
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology.
  The UTAUT2 questionnaire contains 25 questions and evaluates variables including Performance Expectancy, Effort Expectancy, Social Influence, Facility Conditions.
  Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
  Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SACCO, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No